CLINICAL TRIAL: NCT06567171
Title: How Well Ethiopian Parents Assess and Manage Their Children's Postoperative Pain: Descriptive Correlational Study
Status: Completed | Type: Observational
Sponsor: Wachemo University (Other)
Responsible Party: Sponsor
Other Study IDs: NEMMCSH-WCU
Record Dates: First submitted 2024-08-12; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Parent; Pain; Ethiopia; Hospital
Keywords: Parents; Pain; Assessment; Management; Ethiopia; Wachemo University
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: This descriptive correlational study was conducted among 102 parents with children aged between 2 and 12 undergoing elective surgical procedures. — This descriptive correlational study was conducted among 102 parents with children aged between 2 and 12 undergoing elective surgical procedures. Parental use of pain relief strategies (PURPS) and parental postoperative pain management (PPPM) tools were used to collect data on the adequacy of knowledge of the use of different pain relief strategies and the skill of parental pain assessment, respectively. We used Spearman's rank correlation coefficient was used to determine the relationships between pain score given by parents and nurses. The statistical tests were performed at a 95% confidence interval and a 5% significance level.

SUMMARY:
This study aims to evaluate the practice of mothers towards the evaluation and management of postoperative children's pain.According to this study, Parents displayed low to moderate levels of knowledge adequacy towards the use of pain relief methods in relation to their children's postoperative pain and pain management, which indicates the need to provide parents with more information regarding their children's postoperative pain management.

DETAILED DESCRIPTION:
Introduction: Acute postoperative pain in children is common. Although mothers care for their children's pain in most cases, it has been noted that mothers have limited knowledge about pain assessment and management of children.

Objectives: This study aims to evaluate the practice of parents towards evaluating and managing postoperative children's pain.

Method: This descriptive correlational study was conducted among 102 parents with children aged between 2 and 12 undergoing elective surgical procedures. Parental use of pain relief strategies (PURPS) and parental postoperative pain management (PPPM) tools were used to collect data on the adequacy of knowledge of using different pain relief strategies and the skill of parental pain assessment, respectively. Investigators used Spearman's rank correlation coefficient to determine the relationships between pain scores given by parents and nurses. The statistical tests were performed at a 95% confidence interval and a 5% significance level.

ELIGIBILITY:
Inclusion Criteria:

* Parents whose children are receiving elective surgical procedures
* age between the ages of two and twelve in year
* The legal parents' fluency in the local language in speaking, writing, and reading,
* lack of a diagnosis of any visual, auditory, sensory, or other illness

Exclusion Criteria:

Children with

* ASA classifications III or IV,
* significant developmental delays,
* chronic illnesses
* premature births,
* underlying chronic pain conditions (e.g., diabetes)
* a medical history of multiple painful experiences (e.g., malignancies)

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Parents whose children are receiving elective surgical procedures and are between the ages of two and twelve were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
To evaluate the quality of parents management of children's pain in postoperative period using observational tools called PURPS (Parental use of pain relief strategy) and PPPM (Parental postoperative pain measure) | Oct, 2023
  An observational tool was used to measure the quality of parental pain management

CONTACTS AND LOCATIONS:
Locations (1):
- Mitiku Desalegn, Hosa’ina, Snnpr, Ethiopia

IPD SHARING:
Plan to Share IPD: No